212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

| | ,, |
|---|---|
| Statistical Analysis Plan | |
| Title: | A Phase III, randomized, double-blind, placebo-<br>controlled multi-country study to demonstrate efficacy<br>of a single dose of unadjuvanted RSV Maternal<br>vaccine, administered IM to pregnant women 18 to 49<br>years of age, for prevention of RSV associated LRTI<br>in their infants up to 6 months of age |
| eTrack study number and<br>Abbreviated Title | 212171 (RSV MAT-009) |
| Scope: | All analyses for the primary and secondary objectives of the study. Analysis details for tertiary objectives may be described in an SAP Amendment. |
| Date of Statistical Analysis<br>Plan | Amendment 5 Final: 21 Sep 2023 |

APP 9000058193 Statistical Analysis Plan Template V5 (Effective date: 1July2020)

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

## **TABLE OF CONTENTS**

| | | | | | PAGE |
|---|---|---|---|---|---|
| LIS | T OF A | BBREVIA | TIONS | | 7 |
| 1. | DOCU | IMENT H | STORY | | 8 |
| 2. | OBJE | CTIVES/I | NDPOINTS | | q |
| 3. | STUD | Y DESIG | V | | 13 |
| 4. | | | | | |
| | 4.1. | | | | |
| | 4.2. | | | from Analysis Sets | |
| | | 4.2.1. | | Exposed Set (ES) | 24 |
| | | 4.2.2. | Elimination from N | Modified Full Analysis Set for Efficacy | |
| | | | | | 24 |
| | | | | ed Infants from Modified Full Analysis | |
| | | | | Efficacy | |
| | | 4.2.3. | | full Analysis Set for Efficacy (FAS-E) | 24 |
| | | | | ed Infants from Full Analysis Set for | |
| | | | Efficac | y | 24 |
| | | 4.2.4. | Elimination from F | Per protocol analysis set for Efficacy | |
| | | | | | 25 |
| | | | 4.2.4.1. Exclud | ed Infants from Per protocol analysis set | |
| | | | for Effi | cacy (PPS-E) | 25 |
| | | 4.2.5. | Elimination from F | Per-protocol analysis Set for<br>PPS-I) | |
| | | | Immunogenicity (I | PPS-I) | 26 |
| | | | 4.2.5.1. Exclud | ed participants from Per-protocol | |
| | | | | is set for immunogenicity of maternal | |
| | | | | oants | 26 |
| | | | | ed participants from Per-protocol | |
| | | | | ogenicity (PPS-I) analysis set of infant | |
| | | | | pants | 28 |
| | | 4.2.6. | | olicited safety set | |
| | | | | ed participants from Solicited safety set | |
| 5. | STATI | STICAL | NALYSES | | 30 |
| | 5.1. | Demogr | aphy | | 30 |
| | | 5.1.1. | | graphics/baseline characteristics planned | |
| | | | | , | 30 |
| | | 5.1.2. | | erations | |
| | 5.2. | | | | |
| | · | 5.2.1. | | y efficacy endpoints planned in the | |
| | | 0.2 | | | 31 |
| | | | | vity Analyses | |
| | | 5.2.2. | | dary efficacy endpoints planned in the | |
| | | J | protocol | | 33 |
| | 5.3. | Immuno | | | |
| | 0.0. | 5.3.1. | Analysis of immur | nogenicity planned in the protocol | 36 |
| | | 5.3.2. | | erations | |
| | | J.U.Z. | | vity analysis | |
| | | | OOHGILI | * 1. * , GO 1 GO 1 GO 1 GO 1 GO 1 GO 1 GO 1 GO | |

212171 (RSV MAT-009)

| | | | | Statistical Analysis Plan Amend | |
|---|---|---|---|---|---|
| | | | 5.3.2.2. | | |
| | 5.4. | • | | nd reactogenicity | 38 |
| | | 5.4.1. | | of safety and reactogenicity planned in the | 00 |
| | | E 4 0 | | l appoid a rations | |
| | | 5.4.2. | 5.4.2.1. | considerations | |
| | | | 5.4.2.1.<br>5.4.2.2. | Analysis of solicited events Exclusion of implausible solicited Event | |
| | | | 5.4.2.3. | Analysis of Unsolicited Adverse Events | |
| | | | 5.4.2.4. | Combined Solicited and Unsolicited Adverse | 42 |
| | | | 0.4.2.4. | Events | 42 |
| | | | 5.4.2.5. | Other analysis | |
| | | | 0.1.2.0. | Curor analysis | 12 |
| 6. | ANAL | YSIS INT | ERPRETAT | ΓΙΟΝ | 43 |
| 7. | CONE | OUCT OF | ANALYSES | S | 43 |
| | 7.1. | | | ses | |
| | 7.2. | | | ations for interim analyses | |
| | | | | • | |
| 8. | CHAN | IGES FRO | OM PLANN | ED ANALYSES | 44 |
| 9. | NON | CTANDAI | | DERIVATION RULES AND STATISTICAL | |
| 9. | | | | ERIVATION ROLES AND STATISTICAL | 11 |
| | 9.1. | | | vaccination | |
| | 9.2. | | | vaccination | |
| | 3.2. | 9.2.1. | | -offs | |
| | | 0.2.1. | 9.2.1.1. | Assay cut-offs for serology results | |
| | | | 0.2.1.1. | 9.2.1.1.1. Assay cut-offs for central nasal | |
| | | | | swabs | 45 |
| | | 9.2.2. | RTI and L | RTI | |
| | | | 9.2.2.1. | Alternative LRTI / Severe LRTI case definitions | |
| | | | | for data analysis in infants | 47 |
| | | 9.2.3. | Hematolo | gy and Biochemistry parameters | 47 |
| | 9.3. | Statistic | al Method | | 48 |
| 4.0 | | VE0 | | | 40 |
| 10. | | | | Annaland data daminations and statistical models do | |
| | 10.1. | | | standard data derivations and statistical methods | |
| | | 10.1.1. | 10.1.1.1. | of missing data<br>Dates | |
| | | | | Laboratory data | |
| | | | 10.1.1.2. | | |
| | | | 10.1.1.0. | 10.1.1.3.1. Studies with electronic diaries | |
| | | | 10.1.1.4. | Unsolicited adverse events | |
| | | 10.1.2. | | /ation | |
| | | | 10.1.2.1. | Age at vaccination in days | |
| | | | 10.1.2.2. | Age at vaccination in months | |
| | | | 10.1.2.3. | Age at vaccination in years | |
| | | | 10.1.2.4. | Weight | |
| | | | 10.1.2.5. | Height/Length | 50 |
| | | | 10.1.2.6. | Body mass index (BMI) | 50 |
| | | | 10.1.2.7. | Temperature | |
| | | | 10.1.2.8. | Numerical serology results | 50 |

## 212171 (RSV MAT-009) Analysis Plan Amendment 5

| | | | Statistical Analysis Plan Amend | ment 5 |
|---|---|---|---|---|
| | | 10.1.2.9. | Geometric mean titres (GMTs) and | |
| | | | concentrations (GMCs) | 50 |
| | | 10.1.2.10. | Onset day | 51 |
| | | 10.1.2.11. | Duration of events | 51 |
| | | 10.1.2.12. | Counting rules for combining solicited and | |
| | | | unsolicited adverse events | 51 |
| | | 10.1.2.13. | Counting rules for occurrences of solicited | |
| | | | adverse events | |
| | 10.1.3. | Display of | decimals | 51 |
| | | 10.1.3.1. | Percentages | 51 |
| | | | Differences in percentages | |
| | | 10.1.3.3. | Demographic/baseline characteristics statistics | 52 |
| | | 10.1.3.4. | Serological summary statistics | 52 |
| | 10.1.4. | Statistical | methodology | 53 |
| | | 10.1.4.1. | Exact confidence intervals around proportions | 53 |
| | | 10.1.4.2. | Standardized asymptotic confidence intervals | |
| | | | around differences in proportions | 53 |
| | | 10.1.4.3. | Adjusted GMT or GMC ratios | 53 |
| 10.2 | 2. TFL TO | C | | 53 |
| 11 RFI | FERENCES | | | 54 |
| | | | | 0 1 |

## 212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

## **LIST OF TABLES**

| | | PAGE |
|---|---|---|
| Table 1 | Study objectives and endpoints | 9 |
| Table 2 | Study groups, sub-cohorts, interventions, and blinding foreseen in the study: Stage A | 16 |
| Table 3 | Study groups, sub-cohorts, interventions, and blinding foreseen in the study: Stage B | 17 |
| Table 4 | Maternal Participants | 18 |
| Table 5 | Infant participants | 18 |
| Table 6 | Overview of analysis sets and exclusion codes | 19 |
| Table 7 | Elimination code and condition for maternal participants | 26 |
| Table 8 | Elimination code and condition for infant participants | 28 |
| Table 9 | Intensity scales for solicited symptoms in adults | 41 |
| Table 10 | Implausible Solicited Events | 42 |
| Table 11 | MA-RTI case definitions for data analysis in maternal participants | 46 |
| Table 12 | RTI/LRTI case definitions for data analysis in infants | 46 |
| Table 13 | Alternative LRTI / Severe LRTI case definitions in infants | 47 |

## 212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

## **LIST OF FIGURES**

| | | PAGE |
|----------|-----------------------------------------------|------|
| Figure 1 | Study design overview – maternal participants | 13 |
| Figure 2 | Study design overview – infant participants | 14 |

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

## LIST OF ABBREVIATIONS

AE Adverse event

AESI Adverse Events of Special Interest

ANOVA Analysis of Variance
CI Confidence Interval

CRF Case Report Form

CTRS Clinical Trial Registry Summary

eCRF Electronic Case Report Form

ES Exposed Set

FAS Full Analysis Set

GMC Geometric mean antibody concentration

GMT Geometric mean antibody titre

GSK GlaxoSmithKline

HIC High Income Countries

IDMC Independent Data Monitoring Committee

LL Lower Limit of the confidence interval

LLOQ Lower Limit of Quantification

LMIC Low-middle Income Countries

LRTI Lower Respiratory Tract Illness

MAE Medically attended adverse event

MedDRA Medical Dictionary for Regulatory Activities

NA Not Applicable

NB Newborn

PD Protocol Deviation

PPS Per-Protocol Set

RTI Respiratory Tract Illness

SAE Serious Adverse Event

SAP Statistical Analysis Plan

SBIR GSK Biological's Internet Randomization System

SD Standard Deviation

SDTM Study Data Tabulation Model

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

# 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|-------------|-------------|---------------------|
| 02 Nov 2020 | Final | Amendment 1: 05 Oct |
| | | 2020 |
| 01 Nov 2021 | Amendment 1 | Amendment 2: 23 |
| | | Jun 2021 |
| 17 Nov.2022 | Amendment 2 | Amendment 4: 15 |
| | | Mar 2022 |
| 03 Jan 2023 | Amendment 3 | Amendment 4: 15 |
| | | Mar 2022 |
| 09 Mar 2023 | Amendment 4 | Amendment 5: 23 |
| | | Feb 2023 |
| 21 Sep 2023 | Amendment 5 | Amendment 5: 23 |
| - | | Feb 2023 |

# 2. OBJECTIVES/ENDPOINTS

# Table 1 Study objectives and endpoints

| Primary objectives | Primary endpoints |
|---|---|
| To assess the efficacy of a single dose of the RSV Maternal vaccine administered to maternal participants in preventing <i>medically assessed</i> <sup>1</sup> , RSV-associated severe LRTIs in their infant <sup>3</sup> participants up to 6 months of age | From birth (Visit 1-NB) to 6 months (Visit 4-NB), occurrences of medically assessed 1, RSV-associated severe LRTIs according to the case definitions <sup>2</sup> . |
| | OR |
| To assess the efficacy of a single dose of the RSV Maternal vaccine administered to maternal participants in preventing <i>medically assessed</i> <sup>1</sup> , RSV-associated LRTIs of any severity in their infant <sup>3</sup> participants up to 6 months of age | From birth (Visit 1-NB) to 6 months (Visit 4-NB), occurrences of any <i>medically assessed</i> <sup>1</sup> , RSV-associated LRTIs according to the case definitions <sup>2</sup> . |
| | AND |
| To evaluate the safety of the RSV Maternal vaccine in infants born to mothers who were | Occurrence of SAEs, AEs leading to study termination and medically attended AEs from birth up to 6 months after birth <sup>5</sup> . |
| vaccinated with a single IM dose of study vaccine, up to 12 months after birth. | Occurrence of SAEs, AEs leading to study termination and medically attended AEs from birth up to 12 months after birth <sup>5</sup> . |
| Secondary efficacy objectives | Secondary efficacy endpoints |
| To assess the efficacy of a single dose of the RSV Maternal vaccine administered to maternal participants in preventing RSV-associated hospitalization in their infant <sup>3</sup> participants up to 6 months of age. | From birth (Visit 1-NB) to 6 months (Visit 4-NB), occurrences of RSV-associated hospitalizations according to the case definitions <sup>2</sup> . |
| To assess the efficacy of a single dose of the RSV Maternal vaccine administered to maternal participants in preventing, in their infant <sup>3</sup> participants up to 6 months of age, all cause LRTI | From birth (Visit 1-NB) to 6 months (Visit 4-NB), occurrences of all-cause LRTI. |
| To assess the efficacy of a single dose of the RSV Maternal vaccine administered to maternal participants in preventing, in their infant <sup>3</sup> participants up to 6 months of age, all cause LRTI with hospitalization. | From birth (Visit 1-NB) to 6 months (Visit 4-NB), occurrences of all-cause LRTI with hospitalization. |
| To assess the efficacy of a single dose of the RSV Maternal vaccine administered to maternal participants in preventing medically assessed <sup>1</sup> , RSV-associated severe LRTIs in their infant <sup>3</sup> participants up to 12 months of age. | From birth (Visit 1-NB) to 12 months (Visit 5-NB), occurrences of medically assessed, RSV-associated severe (including very severe) LRTIs according to the case definitions <sup>2</sup> . |
| To assess the efficacy of a single dose of the RSV Maternal vaccine administered to maternal participants in preventing medically assessed <sup>1</sup> , RSV-associated LRTIs of any severity in their infant <sup>3</sup> participants up to 12 months of age. | From birth (Visit 1-NB) to 12 months (Visit 5-NB), occurrences of any medically assessed, RSV-associated LRTIs according to the case definitions <sup>2</sup> . |
| To assess the efficacy of a single dose of the RSV Maternal vaccine administered to maternal participants in preventing severe medically assessed <sup>1</sup> , RSV-associated LRTIs for each RSV | From birth (Visit 1-NB) to 6 months (Visit 4-NB), occurrences of severe medically assessed <sup>1</sup> , RSV-associated LRTIs according to the case definition <sup>2</sup> , for RSV subtype A and RSV subtype B separately. |

## 212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

| Statistical Arialysis Plan Amendment 5 |
|---|
| From birth (Visit 1-NB) to 6 months (Visit 4-NB), occurrences of any medically assessed <sup>1</sup> , RSV-associated LRTIs according to the case definition <sup>2</sup> , for RSV subtype A and RSV subtype B separately. |
| From birth (Visit 1-NB) to 4 months (Visit 3-NB), occurrences of severe medically assessed <sup>1</sup> , RSV-associated LRTIs according to the case definitions <sup>2</sup> . |
| From birth (Visit 1-NB) to 4 months (Visit 3-NB), occurrences of any medically assessed <sup>1</sup> , RSV-associated LRTIs according to the case definitions <sup>2</sup> |
| From birth (Visit 1-NB) to 6 months (Visit 4-NB), occurrences of all-cause pneumonia. |
| From birth (Visit 1-NB) to 12 months (Visit 5-NB), occurrences of RSV-associated hospitalizations according to the case definitions <sup>2</sup> . |
| From study intervention administration (Visit 1) to 6 months post-delivery (Contact 1), occurrence of RSV-associated medically attended RTIs (RSV-MA-RTIs) <sup>2</sup> . |
| Secondary immunogenicity endpoints |
| Neutralizing antibody titers against RSV-A |
| Measured on blood samples collected at Day 1 before the study intervention (Visit 1), at Day 31 (Visit 2), and at delivery (Visit 3). |
| Neutralizing antibody titers against RSV-A. |
| Measured on the cord blood sample collected at delivery, or on a blood sample collected from the infant within 72 hours after birth (if no cord blood sample can be obtained) |
| Measured on a blood sample collected at Day 43 (Visit 2-NB), Day 121 (Visit 3-NB), or Day 181 (Visit 4-NB) after birth in 3 sub-cohorts of infants. |
| Infants born to women in the immunogenicity sub-cohort will be randomly assigned (1:1:1) to sample collection at 1 of the 3 timepoints noted. |

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

| | Statistical Analysis Plan Amendment 5 |
|---|---|
| To evaluate the transfer of RSV-specific antibodies from a sub-cohort of maternal participants vaccinated with a single IM dose of the RSV Maternal vaccine to their infants at the | RSVPreF3 IgG-specific antibody concentration measured on blood samples collected at Delivery and cord blood* |
| time of delivery. | The ratio between cord blood* and maternal RSVPreF3 lgG-specific antibody concentrations |
| | * or an infant blood sample collected within 72 hours after birth (if no cord blood sample can be obtained). |
| Secondary safety objectives | Secondary safety endpoints |
| To evaluate reactogenicity of a single IM dose of the RSV Maternal vaccine in stage A maternal participants, during a 7 day follow up period after the study intervention. To evaluate the safety of a single IM dose of the RSV Maternal vaccine in all maternal participants, during a 30 day follow up period after the study | Occurrence of solicited administration site and systemic events in stage A maternal participants, during a 7-day follow-up period after the study intervention (i.e. the day of the intervention and 6 subsequent days). Occurrence of unsolicited adverse events (AEs) in all maternal participants during a 30-day follow-up period after the study intervention (i.e. the day of the intervention and 29 subsequent |
| intervention. To evaluate the safety of a single IM dose of the RSV Maternal vaccine in all maternal participants, from Visit 1 up to 6 months after delivery | days). Occurrence of serious adverse events (SAEs) 5, AEs leading to study termination, and medically attended RTIs in all maternal participants from Visit 1 (Day 1) up to 6 months after delivery. Occurrence of all other medically attended AEs in all maternal participants from Visit 1 (Day 1) up to Day 42 after delivery. |
| To evaluate pregnancy outcomes and pregnancy-related adverse events of special interest after a single IM dose of the RSV Maternal vaccine administered to maternal participants, from Visit 1 up to 6 weeks after delivery (Visit 4). | Pregnancy outcomes <sup>5</sup> from Day 1 (Visit 1) up to 6 weeks after delivery (Day 43 post-delivery, Visit 4). These include live birth with no congenital anomalies, live birth with minor congenital anomaly(ies) only; live birth with at least one major congenital anomaly, fetal death/still birth (antepartum or intrapartum) with no congenital anomalies, fetal death/still birth (antepartum or intrapartum) with only minor congenital anomalies, fetal death/still birth (antepartum or intrapartum) with at least 1 major congenital anomaly; elective/therapeutic termination with no congenital anomalies; elective/therapeutic termination with only minor congenital anomalies, and elective/therapeutic termination with at least 1 major congenital anomaly. |
| | Pregnancy-related adverse events (AEs) of special interest from Day 1 (Visit 1) up to 6 weeks after delivery (Day 43 post-delivery, Visit 4). These include maternal death, hypertensive disorders of pregnancy (gestational hypertension, preeclampsia, pre-eclampsia with severe features including eclampsia), fetal growth restriction, pathways to preterm birth (premature preterm rupture of membranes, preterm labor, provider-initiated preterm birth), gestational diabetes mellitus, chorioamnionitis. 4,5 |
| To evaluate the occurrence of neonatal AEs of special interest (reported up to 6 weeks after birth), in infants born to mothers who were vaccinated with a single IM dose of the RSV Maternal vaccine | The occurrence of neonatal AEs of special interest (reported up to 6 weeks after birth). These include small for gestational age, low birth weight including very low and extremely low birth weight (<2500 g, <1500g, <1000g), congenital anomalies (major external structural defects, internal structural defects, functional defects), neonatal death (in an extremely preterm birth [22≤GA<28 weeks], in a preterm live birth [28≤GA<37 weeks], or in a term live birth), preterm birth. 4.5 |

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5



<sup>1</sup>By "medically assessed" it is meant that the infant was evaluated by a healthcare professional (physician, nurse, etc) for the lower respiratory tract illness.

<sup>2</sup>Case definitions for *RSV-associated medically attended RTIs*, RSV associated LRTIs, surveillance for potential LRTIs, are briefly summarized in Section 9.2.2.

<sup>3</sup>An infant is defined as a child younger than 1 year of age; a neonate is defined as an infant 28 days old or less.

<sup>4</sup>Maternal and neonatal AESI and pregnancy outcomes should be recorded in the eCRF along with assessment of level of diagnostic certainty by GAIA definitions when applicable. Of note, some events of interest fall under a single category but have multiple subcategories. For example, hypertensive disorder of pregnancy is an event with three subcategories that include: 1) gestational hypertension; 2) pre-eclampsia; and 3) pre-eclampsia with severe features (including eclampsia). For each event, the investigator should identify the event and select the applicable sub-category.

<sup>5</sup>The following adverse events are listed by GAIA as events of interest, but will not, for purposes of this study, be reported as AESIs. If any of these events meets the definition for an SAE, the event should be reported as such in the eCRF and the SAE narrative should contain enough information to permit assessment of level of diagnostic certainty by GAIA criteria:

- Pregnancy-related: antenatal bleeding (morbidly adherent placenta, placental abruption, cesarean scar
  pregnancy, uterine rupture), postpartum hemorrhage, non-reassuring fetal status, oligohydramnios,
  polyhydramnios, gestational liver disease (intrahepatic cholestasis of pregnancy, acute fatty liver of pregnancy),
  maternal sepsis.
- Neonatal: neonatal encephalopathy, congenital microcephaly (postnatally or prenatally diagnosed), neonatal
  infections (blood stream infections, meningitis, respiratory infection), respiratory distress in the neonate, failure to
  thrive, large for gestational age, macrosomia.

## STUDY DESIGN

### Figure 1 Study design overview – maternal participants



GA = Gestational age; I = immune response; (S)AE = (serious) adverse event; RTI = respiratory tract illness Visit 2 may be replaced by Visit 3 in case of premature delivery.

All = all participants

Refer to Protocol Amendment 5 Section 6.3.2 for detailed description of Stage A and Stage B. Refer to Protocol Amendment 5 Section 6.3.2.1.1 for additional description of the Stage A sub-cohort.

Solicited events will be evaluated for all participants in Stage A only

\* Any pregnancy-related event of special interest identified after Visit 4 should also be reported. In addition to the monthly contacts between Visit-2 and the Delivery visit, additional not pre-specified visits and contacts (any desired frequency) can be made between Visit-2 and the Delivery visit, as per investigator's or maternal participant's discretion.

As from protocol Amentment 4, blood samples will be collected at delivery from all maternal participants. Placental samples will be collected at delivery from all maternal participants, if feasible

Due to the stop on study enrolment and vaccination, nasal swab samples will no longer be collected from any maternal participant and no MA-RTI assessment visit will be performed, but the MAEs associated with an RTI will continue to be reported, as applicable.

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

Figure 2 Study design overview – infant participants



I = immune response; (S)AE = (serious) adverse event; RTI = respiratory tract illness Stage A + Stage B – all participants:

\*If cord-blood was not collected at delivery/birth, a blood sample should be collected from the infant within 72 hours post birth. Applies to all participants in Stage A and Stage B.

An additional recommended safety contact may be performed 8-days post-birth if deemed necessary by the investigator or by the parent/LAR(s).

Due to the stop on study enrolment and vaccination, blood samples will no longer be collected at V2-NB, V3-NB or V4-NB.

- Study Type: self-contained
- Study Duration: Approximately 10 to 11 months (including the screening visit) for maternal participants; approximately 1 year after birth for infant participants.
- Blinding is as described in Table 2 and Table 3.
- Randomized intervention allocation: A minimum of 4600 and up to a maximum of 10,000 pregnant women (maternal participants) will be randomly assigned (2:1) to receive the investigational vaccine or control (placebo) at Visit 1. Randomization will take place in 2 sequential stages, A and B. Approximately 4,600 maternal participants will be randomized into Stage A. Stage B will only start after the last participant is randomized in Stage A. Participants in stage A will be randomized (12:2:2:2:6:1:1:1 ratio) to be in the RSV group, in one of the 3 infant blood sampling sub-cohorts and receiving the investigational vaccine (RSVMAT BS1 (Day 43), RSVMAT BS2 (Day 121), RSVMAT BS3 (Day 181)), in the Control group, or in one of the 3 infant blood sampling sub-cohorts receiving placebo (Control BS1 (Day 43), Control\_BS2 (Day 121), Control BS3 (Day 181)). Randomization will be via the automated internet-based system (SBIR). The system's randomisation algorithm of maternal enrolment will use a minimisation procedure accounting for maternal age at the time of the study intervention (18-34, 35-39, >40 years of age), gestational age at the time of the study intervention  $(24^{0/7}-28^{0/7}; 28^{1/7}-34^{0/7})$ , and center. Minimisation factors will have equal weight in the minimisation algorithm.
- Study (intervention) groups are described in Table 2 and Table 3
- Data collection: standardized Electronic Case Report Form (eCRF). E-Diaries will be used to collect solicited event data.

<sup>\*\*</sup>Any Neonatal AE of specific interest identified after Day 43 should also be reported.

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

• Safety monitoring will be conducted by an unblinded Independent Data Monitoring Committee (IDMC) and by an unblinded Safety Review Team\*. The analyses for IDMC safety evaluations will be described in a separate SAP for IDMC.

<sup>\*</sup> Due to the safety signal observed, the study was fully unblinded to ensure the safety of the participants.

Table 2 Study groups, sub-cohorts, interventions, and blinding foreseen in the study: Stage A

Approximately 4,600 maternal participants will be randomized during Stage A.

| | | | | | | | | | Blinding | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Study<br>groups | Maternal pa | ırticipants (M | ) | | | Infant participan | ts (I) | Study Groups<br>for<br>Randomization | M only | M + I | I only |
| | ~Number | Age in<br>Years<br>(Min/Max) | Intervention Maternal Blood Sampling Sub-cohorts | | • | Infant Blood Sampling ( | | (Allocation<br>12:2:2:2:6:1:1:1) | Screen-<br>ing | Up to D181<br>post<br>delivery/birth | D271, D366<br>post<br>delivery/birth |
| | | | | Name | ~Number | Name | ~Number | | - | Double blind | Double blind |
| | | 18-49 | RSV_MAT | RSV_MAT_0 | ~2,040 | RSV_MAT_0 | ~2,040 | RSVMAT_0 | | • | |
| DOV MAT | 2.007 | 18-49 | RSV_MAT | RSV_MAT_I | ~1020 | RSV_MAT_BS1 | ~340 | RSVMAT_BS1 | | • | - |
| RSV_MAT | ~3,067 | | | | | RSV_MAT_BS2 | ~340 | RSVMAT_BS2 | • | • | |
| | | | | | | RSV_MAT_BS3 | ~340 | RSVMAT_BS3 | | • | |
| | | 18-49 | Control | Control_0 | ~1020 | Control_0 | ~1020 | Control_0 | | • | |
| Control | 1 522 | 18-49 | Control | Control_I | ~510 | Control_BS1 | ~170 | Control_BS1 | | • | |
| | ~1,533 | | | | | Control_BS2 | ~170 | Control_BS2 | • | • | • |
| | | | | | | Control_BS3 | ~170 | Control_BS3 | | • | |

Control = Placebo; Infant sub-cohorts are abbreviated "BS1;" "BS2;" BS3" and correspond to visits 2-NB (Day 43), 3-NB (Day 121) and 4-NB (Day 181), respectively.

RSVMAT\_0 and Control\_0 = maternal and infant participants who are not in a sub-cohort for immune response assessment.

 $RSVMAT\_I \ and \ Control\_I = maternal \ sub-cohorts \ for \ immune \ response \ assessment.$ 

RSVMAT\_BS1, \_BS2, \_BS3 = infants born to women in the RSVMAT\_I sub-cohort and evaluated for immune response at the designated timepoint (D43, D121 or D181).

Control\_BS1, \_BS2, \_BS3 = infants born to women in the Control\_I sub-cohort evaluated for immune response at the designated timepoint (D43, D121 or D181).

21 Sep 2023 

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

## Table 3 Study groups, sub-cohorts, interventions, and blinding foreseen in the study: Stage B

Approximately a maximum of 5,400 maternal participants may be randomized during Stage B.

Stage B will only start after the last participant is randomized in Stage A.

| | | Age of maternal<br>participant at enrolment<br>(Min/Max) | | | Blinding | | |
|---|---|---|---|---|---|---|---|
| Study groups | Number of<br>maternal<br>participants | | Intervention name | Study groups for randomization (Allocation 2:1) | Maternal<br>participants<br>Only<br>(Screening) | Maternal participants V1-C1 Infant participants V1-NB – V4NB (double-blind) | Infant participants<br>only<br>Contact 2-NB – V5-<br>NB<br>(double blind) |
| RSV_MAT | ~3,600 | 18 – 49 years | RSV_MAT | RSV_MAT | • | • | • |
| Control | ~1,800 | 18 – 49 years | Control | Control | • | • | • |

21 Sep 2023 

## 4. ANALYSIS SETS

## 4.1. Definition

For the purpose of the analysis the following analysis sets are defined.

# Table 4 Maternal Participants

| Analysis Set | Description |
|---|---|
| Enrolled | All maternal participants who completed the informed consent process and signed the informed consent form. |
| Exposed | All maternal participants who received the study intervention. The allocation in a group is done in function of the administered intervention. |
| Per Protocol -<br>Immunogenicity | All maternal participants who received the study intervention to which they were randomised and have post-vaccination data minus participants with protocol deviations that lead to exclusion. |
| Solicited Safety –<br>Stage A only | All maternal participants in the Exposed Set who have solicited safety data |

## Table 5 Infant participants

| Analysis Set | Description |
|---|---|
| Exposed | Infants live-born to exposed maternal participants, whose parents/LARs completed the |
| | informed consent process and signed the informed consent form. |
| Per Protocol - | All infant participants in the Exposed set minus those who (a) were born less than 4 weeks |
| Immunogenicity | post- maternal participant vaccination and/ or (b) have protocol deviations that lead to |
| | exclusion. |
| Full Analysis - | All infant participants in the Exposed set. |
| Efficacy | |
| Modified Full | All infant participants in the Exposed set who were born after at least 4 weeks of |
| Analysis - Efficacy | vaccination. |
| Per Protocol - | All infant participants in the Modified Full Analysis – Efficacy set minus those who have |
| Efficacy | protocol deviations that lead to exclusion. |

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

Table 6 Overview of analysis sets and exclusion codes

| | Code | Description | | Maternal | analysis s | et | | | Infant analysi | is set | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Determined in mother or infant | | | Enrolled | Exposed | Per Protocol -<br>Immunogenicity | Solicited Safety | Exposed | Per Protocol -<br>Immunogenicity | Modified Full<br>Analysis -<br>Efficacy | Full Analysis -<br>Efficacy | Per Protocol -<br>Efficacy |
| Mother | 800, 800# | Fraudulent Data | Υ | Υ | Υ | Υ | Υ | Υ | Υ | Υ | Υ |
| Mother | 900, 900# | Invalid informed consent | Υ | Υ | Υ | Υ | Υ | Υ | Υ | Υ | Υ |
| Mother | 1030, 1030# | Study vaccine not administered | | Y | Y | Y | Y | Y | Υ | Y | Y |
| Mother | 1040.Vx+*,<br>1040# | Administration of concomitant vaccine(s) forbidden in the protocol | | | Υ | | | Y | | | Y |
| Mother | 1050, 1050# | Randomisation failure | | | Υ | | | Υ | | | Υ |
| Mother | 1060, 1060# | Randomisation code was brokena | | | Y | | | Υ | | | Υ |
| Mother | 1070, 1070# | Mother got vaccinated with the correct vaccine but incorrect volume | | | Y | | | Υ | | | Y |
| Mother | 1070, 1070# | Vaccination not according to protocol (site of injection, route of administration, wrong replacement of study treatment administered) | | | Y | | | Y | | | Y |
| Mother | 1070, 1070# | Study treatment not prepared as per protocol (e.g. reconstitution) | | | Y | | | Y | | | Y |
| Mother | 1070, 1070# | Other deviations related to wrong study treatment/ administration/dose | | | Υ | | | Y | | | Y |

21 Sep 2023 

## 212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

| | Code | Description | | Maternal | analysis s | et | | | Infant analysi | is set | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Determined in mother or infant | | | Enrolled | Exposed | Per Protocol - | Solicited Safety | Exposed | Per Protocol -<br>Immunogenicity | Modified Full<br>Analysis -<br>Efficacy | Full Analysis -<br>Efficacy | Per Protocol -<br>Efficacy |
| Mother | 1070, 1070# | Study treatment administered while contraindicated | | | Y | | | Y | | | Y |
| Mother | 1080, 1080# | Vaccine temperature deviation | | | Υ | | | Υ | | | Y |
| Mother | 1090, 1090# | Expired vaccine administered | | | Y | | | Υ | | | Y |
| Mother | 1160 | No post-vaccination solicited safety data- Stage A participants only | | | | Y | | | | | |
| Mother | 2010, 2010# | Protocol violation (inclusion/exclusion criteria) | | | Υ | | | Υ | | | Y |
| Mother | 2040.Vx+*,<br>2040# | Administration of any medication/product forbidden by the protocol | | | Y | | | Υ | | | Υ |
| Mother | 2050.Vx+*,<br>2050# | Intercurrent medical conditions/concomitant medications which are exclusionary as per protocol | | | Y | | | Y | | | Y |
| Mother | 2060.Vx+*,<br>2060# | Concomitant infection related to the vaccine which may influence the immune response | | | Y | | | Y | | | Y |
| Mother | 2070.Vx+*,<br>2070# | Concomitant infection not related to the vaccine but may influence the immune response | | | Y | | | Y | | | Y |

21 Sep 2023 

## 212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

| | Code | Description | | Maternal | analysis s | et | | | Infant analys | is set | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Determined in mother or infant | | | Enrolled | Exposed | Per Protocol -<br>Immunogenicity | Solicited Safety | Exposed | Per Protocol -<br>Immunogenicity | Modified Full<br>Analysis -<br>Efficacy | Full Analysis -<br>Efficacy | Per Protocol -<br>Efficacy |
| Mother | 2090.Vx | Participant did not comply with blood sample schedule | | _ | Y | | | | | | |
| Mother | 2100.Vx | Serology result not available (immunogenicity sample collected but invalid/no result) | | | Y | | | | | | |
| Mother | 2120.Vx | Obvious incoherence or abnormality or error in the data | | | Y | | | | | | |
| Mother | 2130.Vx | Testing performed on serology samples not aligned with ICF | | | Y | | | | | | |
| Mother | 2110.Vx | Immunogenicity sample collected but GSK decided not to test | | | Y | | | | | | |
| Infant | 800 | Fraudulent Data | | | | | Υ | Υ | Υ | Y | Υ |
| Infant | 900 | Invalid informed consent | | | | | Y* | Υ | Υ | Y | Y |
| Infant | 2010 | Protocol violation (inclusion/exclusion criteria) | | | | | | Y | | | Y |
| Infant | 2050.Vx | Intercurrent medical conditions which are exclusionary as per protocol | | | | | | Y | | | Y |
| Infant | 2090.Vx | Participant did not comply with blood sample schedule | | | | | | Y | | | |

21 Sep 2023 

## 212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

| | Code | Description | | Maternal | analysis s | et | | | Infant analysi | s set | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Determined in mother or infant | | | Enrolled | Exposed | Per Protocol -<br>mmunogenicity | Solicited Safety | Exposed | Per Protocol -<br>Immunogenicity | Modified Full<br>Analysis -<br>Efficacy | Full Analysis -<br>Efficacy | Per Protocol -<br>Efficacy |
| Infant | 2100.Vx | Serology result not available<br>(immunogenicity sample collected<br>but invalid/no result) | | | | | | Y | | | |
| Infant | 2120.Vx | Obvious incoherence or abnormality or error in the data | | | | | | Y | | | |
| Infant | 2130.Vx | Testing performed on serology samples not aligned with ICF | | | | | | Y | | | |
| Infant | 2131.Vx | Testing performed on nasal samples not aligned with ICF | | | | | | | | | Y |
| Infant | 2110.Vx | Immunogenicity sample collected but GSK decided not to test | | | | | | Y | | | |
| Infant | 2040.Vx+,<br>2040# | Administration of any medication/product forbidden by the protocol (leading to elimination from PPS-E and PPS-I) | | | | | | Y | | | Y |
| Infant | 2140Vx+ | Administration of any medication/product forbidden by the protocol (leading to elimination from PPS-I) | | | | | | Y | | | |
| Infant | 2240 | Administration of any medication/product forbidden by the protocol (leading to elimination from PPS-E) | | | | | | | | | Y |

21 Sep 2023 

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

| | Code | Description | | Maternal | analysis s | et | | | Infant analysi | s set | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Determined in<br>mother or<br>infant | | | Enrolled | Exposed | Per Protocol -<br>mmunogenicity | Solicited Safety | Exposed | Per Protocol -<br>mmunogenicity | Modified Full<br>Analysis -<br>Efficacy | Full Analysis -<br>Efficacy | Per Protocol -<br>Efficacy |
| Infant | 2060.Vx,<br>2060# | Concomitant infection related to the vaccine which may influence immune response | | | | | | Y | 2 3 | | Y |
| Infant | 2070.Vx,<br>2070# | Concomitant infection not related to the vaccine but may influence immune response | | | | | | Y | | | Y |
| Infant | 3100 | Birth is less than 4 weeks post-vaccination | | | | | | Y | Υ | | Y |

in case a mother withdraws consent or does not consent for the baby, we still report SAEs/AESIs for the infants if collected

21 Sep 2023 

<sup>.</sup>Vx indicates participants whose data will be eliminated from a specific endpoint/visit

<sup>.</sup>Vx+ indicates participants whose data will be eliminated from a specific endpoint/visit onwards

Y indicates exclusion

<sup>#</sup> Carry forward elimination from mother to infant

<sup>&</sup>lt;sup>a</sup> Randomization code was broken (1060, 1060#) does not apply to the unblinding of all participants during the study due to the stop on study enrollment and vaccination and the study was fully unblinded

## 4.2. Criteria for eliminating data from Analysis Sets



# 4.2.1. Elimination from Exposed Set (ES)



# 4.2.2. Elimination from Modified Full Analysis Set for Efficacy (modified FAS-E)

### 4.2.2.1. Excluded Infants from Modified Full Analysis Set for Efficacy

An infant will be excluded from the modified FAS efficacy analysis under the following conditions:

| Code | Condition under which the code | Visit (timepoints) where the code is |
|---|---|---|
| | is used | applicable |
| 800, 800# | Fraudulent data | All |
| 900, 900# | Invalid informed consent | All |
| 1030# | Study vaccine not administered | All |
| 3100 | Birth is less than 4 weeks post-vaccination | All |

<sup>#</sup> Carry forward elimination from mother to infant

## 4.2.3. Elimination from Full Analysis Set for Efficacy (FAS-E)

### 4.2.3.1. Excluded Infants from Full Analysis Set for Efficacy

An infant will be excluded from the FAS efficacy analysis under the following conditions:

| Code | Condition under which the code is | Visit (timepoints) where the code is |
|---|---|---|
| | used | applicable |
| 800, 800# | Fraudulent data | All |
| 900, 900# | Invalid informed consent | All |
| 1030# | Study vaccine not administered | All |

<sup>#</sup> Carry forward elimination from mother to infant

## 4.2.4. Elimination from Per protocol analysis set for Efficacy (PPS-E)

## 4.2.4.1. Excluded Infants from Per protocol analysis set for Efficacy (PPS-E)

A participant will be excluded from the PPS efficacy analysis under following conditions:

| Code | Condition under which the code is used | Visit (timepoints) where the code is applicable |
|---|---|---|
| 800, 800# | Fraudulent data | All |
| 900, 900# | Invalid informed consent | All |
| 1030# | Study vaccine not administered | All |
| 3100 | Birth/Delivery is less than 4 weeks post-vaccination | All |
| 1040# | Administration of concomitant vaccine(s) forbidden in the protocol | All |
| 1050# | Randomisation failure | All |
| 1060# | Randomisation code was broken | All |
| 1070# | Mother got vaccinated with the correct vaccine but containing an incorrect volume | All |
| 1070# | Vaccination not according to protocol (site of injection, route of administration, wrong replacement of study treatment administered) | All |
| 1070# | Study treatment not prepared as per protocol (e.g. reconstitution) | All |
| 1070# | Other deviations related to wrong study treatment/administration/dose | All |
| 1070# | Study treatment administered while contraindicated | All |
| 1080# | Vaccine temperature deviation | All |
| 1090# | Expired vaccine administered | All |
| 2010,<br>2010# | Protocol violation (inclusion/exclusion criteria) | All |
| 2040* | Administration of any medication/product forbidden by the protocol (leading to elimination from PPS-E and PPS-I) | All |
| 2240* | Administration of any medication/product forbidden by the protocol (leading to elimination from PPS-E) | All |
| 2040* | Administration of any medication/product forbidden by the protocol (leading to elimination from PPS-E and PPS-I) | All |
| 2050.Vx* | Intercurrent medical conditions/concomitant medications which are exclusionary as per protocol | All |

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

| Code | Condition under which the code is used | Visit (timepoints) where the code is applicable |
|---|---|---|
| 2050#* | Maternal intercurrent medical conditions which are exclusionary as per protocol | All |
| 2060#*<br>2060* | Concomitant infection related to the vaccine which may influence immune response | All |
| 2070#*<br>2070* | Concomitant infection not related to the vaccine but may influence immune response | All |
| 2120.Vx | Obvious incoherence or abnormality or error in data | All |
| 2131.Vx | Testing performed on nasal samples not aligned with ICF | All |

<sup>.</sup>Vx indicates participants whose efficacy data will be eliminated from a specific endpoint

# 4.2.5. Elimination from Per-protocol analysis Set for Immunogenicity (PPS-I)

# 4.2.5.1. Excluded participants from Per-protocol analysis set for immunogenicity of maternal participants

A participant will be excluded from the PPS immunogenicity analysis under the following conditions:

 Table 7
 Elimination code and condition for maternal participants

| Code | Condition under which the code is used | Visit (timepoints) where the code is applicable |
|---|---|---|
| 800 | Fraudulent data | All |
| 900 | Invalid informed consent | All |
| 1030 | Study vaccine not administered | All |
| 1040.Vx+* | Administration of concomitant | All |
| | vaccine(s) forbidden in the protocol | |
| 1050 | Randomisation failure | All |
| 1060 | Randomisation code was broken | All |
| 1070* | Mother got vaccinated with the | All |
| | correct vaccine but incorrect volume | |
| 1070* | Vaccination not according to | All |
| | protocol (site of injection, route of | |
| | administration, wrong replacement | |
| | of study treatment administered) | |
| 1070* | Study treatment not prepared as per | All |
| | protocol (e.g. reconstitution) | |
| 1070* | Other deviations related to wrong | All |
| | study treatment/administration/dose | |

<sup>#</sup> Carry forward elimination from mother to infant

<sup>\*</sup> Attribution of these elimination codes to participant need CRDL review of individual listing

## 212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

| | T | Statistical Analysis Flan Americanent 5 |
|---|---|---|
| Code | Condition under which the code is | Visit (timepoints) where the code |
| | used | is applicable |
| 1070* | Study treatment administered while | All |
| 10/0 | contraindicated | 7 111 |
| 1000 | | A 11 |
| 1080 | Vaccine temperature deviation | All |
| 1090 | Expired vaccine administered | All |
| 2010 | Protocol violation | All |
| | (inclusion/exclusion criteria) | |
| 2040.Vx+* | Administration of any | Visit 2/Day 31, |
| | medication/product forbidden by the | Visit 3/Delivery |
| | protocol | |
| 2050.Vx+* | Intercurrent medical conditions | Visit 2/Day 31, |
| | which are exclusionary as per | Visit 3/Delivery |
| | protocol | |
| 2060.Vx+* | Concomitant infection related to the | Visit 2/Day 31, |
| 2000. VX | vaccine which may influence | Visit 3/Delivery |
| | immune response | Tion Si Don't Or y |
| 2070.Vx+* | Concomitant infection not related to | Visit 2/Day 31, |
| 20/0.VX | | Visit 2/Day 31,<br>Visit 3/Delivery |
| | the vaccine but may influence | Visit 3/Delivery |
| 2000 17 | immune response | V' '- 2/D 21 |
| 2090.Vx | Participants did not comply with | Visit 2/Day 31, |
| | blood sample schedule: | Visit 3/Delivery |
| | • For PPS at Visit 2/Day 31, | |
| | check the interval from | |
| | vaccination to day 31 | |
| | BS = -10/+15 days; | |
| | DS 10/+15 days, | |
| | • For PPS at Visit 3/Delivery, | |
| | check the interval from delivery | |
| | to delivery $BS = -1/+3$ days | |
| 2100.Vx | Serological results not available | Visit 1/Day 1 |
| | (immunogenicity sample collected but | Visit 2/Day 31, |
| | invalid/no result) | Visit 3/Delivery |
| 2120.Vx | Obvious incoherence or abnormality | Visit 2/Day 31, |
| 2120. 7 A | or error in the data | Visit 3/Delivery |
| | or error in the data | VISIC SI DOM VOI Y |
| 2130.Vx | Testing performed on serology | Visit 2/Day 31, |
| | samples not aligned with ICF | Visit 3/Delivery |
| 211037 | 1 0 | · |
| 2110.Vx | Immunogenicity sample collected | Visit 1/Day 1 |
| | but GSK decided not to test | Visit 2/Day 31, |
| | | Visit 3/Delivery |

Attribution of these elimination codes to participant need CRDL review of individual listing

<sup>.</sup>Vx+ indicates participants whose immunogenicity data will be eliminated from a specific visit onwards;

<sup>.</sup>Vx indicates participants whose immunogenicity data will be eliminated from a specific visit.

212171 (RSV MAT-009)

## Statistical Analysis Plan Amendment 5

# 4.2.5.2. Excluded participants from Per-protocol immunogenicity (PPS-I) analysis set of infant participants

An infant participant will be excluded from the PPS immunogenicity analysis under following conditions:

 Table 8
 Elimination code and condition for infant participants

| Code | Condition under which the code is used | Visit (timepoints) where the |
|---|---|---|
| 800, 800# | Fraudulent data | code is applicable All |
| 900, 900# | Invalid informed consent | All |
| 1030# | Study vaccine not administered | All |
| 1030#<br>1040.Vx#+* | Administration of concomitant | All |
| 1040. V X#+** | | All |
| 1050# | vaccine(s) forbidden in the protocol Randomisation failure | A 11 |
| 1050# | | All |
| 1060# | Randomisation code was broken | All |
| 1070#* | Mother got vaccinated with the | All |
| 4.0 = 0.114 | correct vaccine but incorrect volume | |
| 1070#* | Vaccination not according to | All |
| | protocol (site of injection, route of | |
| | administration, wrong replacement | |
| 10-000 | of study treatment administered) | |
| 1070#* | Study treatment not prepared as per | All |
| | protocol (e.g. reconstitution) | |
| 1070#* | Other deviations related to wrong | All |
| | study treatment/administration/dose | |
| 1070#* | Study treatment administered while | All |
| | contraindicated | |
| 1080# | Vaccine temperature deviation | All |
| 1090# | Expired vaccine administered | All |
| 2010, 2010# | Protocol violation | All |
| | (inclusion/exclusion criteria) | |
| 2040#* | Administration of any | All |
| | medication/product forbidden by the | |
| | protocol | |
| 2140.#* | Administration of any | All |
| | medication/product forbidden by the | |
| | protocol | |
| 2040Vx* | Administration of any | Visit 1-NB/Birth |
| | medication/product forbidden by the | Visit 2-NB/Day 43 post-birth <sup>a</sup> |
| | protocol | Visit 3-NB/Day 121 post-birth <sup>a</sup> |
| | _ | Visit 4-NB/Day 181 post-birth <sup>a</sup> |
| 2140Vx* | Administration of any | Visit 1-NB/Birth |
| | medication/product forbidden by the | Visit 2-NB/Day 43 post-birth <sup>a</sup> |
| | protocol (leading to elimination | Visit 3-NB/Day 121 post-birth <sup>a</sup> |
| | from PPS-I) | Visit 4-NB/Day 181 post-birth <sup>a</sup> |

## 212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

| | | Statistical Analysis Plan Amendment 5 |
|---|---|---|
| Code | Condition under which the code is | Visit (timepoints) where the |
| | used | code is applicable |
| 2050.Vx#* | Intercurrent medical conditions | All |
| | which are exclusionary as per | |
| | protocol | |
| 2050.Vx* | Intercurrent medical conditions | All |
| | which are exclusionary as per | |
| | protocol | |
| 2060.Vx#+* | Concomitant infection related to the | All |
| 2060.Vx+* | vaccine which may influence | |
| | immune response | |
| 2070.Vx#+* | Concomitant infection not related to | All |
| 2070.Vx+* | the vaccine but may influence | |
| | immune response | |
| 2090.Vx | Participants did not comply with | Visit 1-NB/Birth |
| | blood sample schedule | Visit 2-NB/Day 43 post-birth <sup>a</sup> |
| | • For PPS at Visit 1/Day 1 check | Visit 3-NB/Day 121 post-birth <sup>a</sup> |
| | the interval of day 1 BS -0/+3 | Visit 4-NB/Day 181 post-birth <sup>a</sup> |
| | days; | |
| | • For PPS at Visit 2/Day 43 post- | |
| | birth, check the interval of day | |
| | 43 BS -12/+18 days; | |
| | • For PPS at Visit 3/Day 121 | |
| | post-birth, check the interval of | |
| | day 121 BS -10/+20 days; | |
| | • For PPS at Visit 4/Day 181 | |
| | post-birth, check the interval of | |
| | day 181 -15/+20 days | |
| 2100.Vx | Serological results not available | Visit 1-NB/Birth |
| 2100. V X | (immunogenicity sample collected but | Visit 1-NB/Day 43 post-birth <sup>a</sup> |
| | invalid/no result) | Visit 3-NB/Day 121 post-birth <sup>a</sup> |
| | | Visit 4-NB/Day 181 post-birth <sup>a</sup> |
| 2120.Vx | Obvious incoherence or abnormality | Visit 4-NB/Birth |
| 2120. V A | or error in the data | Visit 2-NB/Day 43 post-birth <sup>a</sup> |
| | of cirol in the data | Visit 3-NB/Day 121 post-birth <sup>a</sup> |
| | | Visit 4-NB/Day 181 post-birth <sup>a</sup> |
| 2130.Vx | Testing performed on serology | Visit 4-NB/Day 181 post-oirtii Visit 1-NB/Birth |
| 4130. V X | samples not aligned with ICF | Visit 1-NB/Birtii Visit 2-NB/Day 43 post-birth <sup>a</sup> |
| | samples not anglied with ICF | Visit 2-NB/Day 43 post-birth <sup>a</sup> |
| | | Visit 4-NB/Day 181 post-birth <sup>a</sup> |
| 2110.Vx | Immunogenicity sample collected | Visit 4-NB/Day 181 post-birth Visit 1-NB/Birth |
| ∠110. V X | but GSK decided not to test | |
| | but GSK decided not to test | Visit 2-NB/Day 43 post-birth <sup>a</sup> |
| | | Visit 3-NB/Day 121 post-birth <sup>a</sup> |
| 2100 | Dight in Lang diagram 4 | Visit 4-NB/Day 181 post-birth <sup>a</sup> |
| 3100 | Birth is less than 4 weeks post- | All |
| | vaccination. | |

Attribution of these elimination codes to participant need CRDL review of individual listing

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

- # Carry forward elimination from mother to infant
- Vx+ indicates participants whose immunogenicity data will be eliminated from a specific visit onwards;
- Vx indicates participants whose immunogenicity data will be eliminated from a specific visit.
- <sup>a</sup> As per Protocol Amendment 4, infant blood samples will not be collected at V2-NB, V3-NB and V4-NB. 2090.Vx, 2100.Vx, 2120.Vx, 2130.Vx will not be applicable to infant participants whose blood samples are not collected under Protocol Amendment 4.

### 4.2.6. Elimination from solicited safety set

### 4.2.6.1. Excluded participants from Solicited safety set

Code 1030 (Study vaccine not administered at all), code 800 (fraudulent data), code 900 (invalid informed consent) and code 1160 (no post-vaccination solicited safety data only for Stage A participants) will be used for identifying participants eliminated from the solicited safety set.

### 5. STATISTICAL ANALYSES

Standard data derivation rules and stat methods are described in section 10.1 while the study specific data derivation rules and stat methods are described in section 9.

## 5.1. Demography

# 5.1.1. Analysis of demographics/baseline characteristics planned in the protocol

These analyses will be performed on the Exposed set (ES) for maternal and infant participants and on the modified Full Analysis - Efficacy set (modified FAS-E) for infant participants. Analysis may also be repeated on the Per Protocol set for immunogenicity for maternal as well as infant participants.

For all maternal participants, demographic characteristics (e.g., age at vaccination (18-34, 35-39,  $\geq$ 40 years of age), gestational age at vaccination (24<sup>0/7</sup> - 28<sup>0/7</sup>, 28<sup>1/7</sup> - 34 <sup>0/7</sup>weeks), geographic ancestry) will be summarized by group and overall using descriptive statistics. The interval in days between maternal vaccination and delivery will be calculated and summarized by group using descriptive statistics.

For their infants, demographic characteristics (e.g., gestational age at time of delivery (≥ 37 weeks; < 37 weeks), sex, weight, length, head circumference, geographic ancestry, apgar score), and lifestyle characteristics (e.g., living environment, household composition, breastfeeding, passive smoking and extent of contact with children less than 6 years of age) will be summarised by group, and for each immunogenicity sub-cohort within each group, using descriptive statistics.

- Frequency tables will be generated for categorical variables such as gestational age at time of delivery ( $\geq$  37 weeks).
- Mean, median, standard deviation and range will be provided for continuous data such as age.

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

Demographics and baseline characteristics as well as the lifestyle characteristics may be reported by geographic region and by economic region (LMIC and HIC).

### 5.1.2. Additional considerations

Demographic characteristics will also be summarized on the Enrolled Set for public disclosure.

Subgroup analysis for demographic characteristics by age category at vaccination (18 – 34, 35-39;  $\geq$  40 years) for maternal participants and by gestational age at birth ( $\geq$  37 weeks or < 37 weeks) for infant participants will also be performed on ES or modified FAS-E for infant participants.

Participants disposition will be summarized by group using descriptive statistics:

- Number of maternal participants enrolled, randomised, vaccinated, eligible for maternal efficacy populations and withdrawn including withdrawal reasons in each group and overall will be tabulated.
- Number of infants enrolled, eligible for infant efficacy populations and withdrawn including withdrawal reasons will be tabulated by group, by sub-cohort within each group and overall.

Vital signs will not be summarized for this study.

Summary of important protocol deviations leading to elimination will be tabulated by group and overall. An individual listing will also be provided.

Summary of medical history will be performed on ES by Medical Dictionary for Regulatory Activities (MedDRA) and preferred term.

## 5.2. Efficacy

# 5.2.1. Analysis of primary efficacy endpoints planned in the protocol

The primary analysis of vaccine efficacy (VE) will be based on the modified Full Analysis - Efficacy set for infants (modified FAS-E). A secondary analysis based on the Full Analysis – Efficacy set (FAS-E) and the Per Protocol - Efficacy set for infants will be performed to complement the modified FAS-E analysis.

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

| | Statistical Analysis Plan Amendment 5 |
|---|---|
| Primary Efficacy Endpoints – Infant participants | Statistical Analysis Methods |
| From birth to 6 months, occurrences of medically assessed, RSV-associated severe LRTIs according to the case definitions. | CCI |
| OR From birth to 6 months, occurrences of any medically assessed, RSV-associated LRTIs according to the case definitions. | |
| CCI | |

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5



### 5.2.1.1. Sensitivity Analyses

Supportive analysis of time to confirmed RSV-LRTI of any severity and time to confirmed severe RSV-LRTI will be conducted by using Kaplan-Meier cumulative incidence curves.

Sub-group analyses by regions and by key demographic characteristics may also be explored. In addition, efficacy analyses stratified by VE reported for geographic regions (North America, Central America & Caribbean, and South America), economic regions (LMIC and HIC), RSV type and RSV seasonality (year-round circulation and seasonal circulation) may be included in the clinical study report.

Supportive analyses on primary efficacy endpoints based on the modified FAS-E will also be conducted for RSV-associated LRTI cases confirmed by central laboratory tests and PCR confirmed local laboratory tests and by all RSV tests (central and all local laboratory tests).

## 5.2.2. Analysis of secondary efficacy endpoints planned in the protocol

The primary analysis of VE on secondary efficacy endpoints in infants will be based on the modified Full Analysis - Efficacy set (modified FAS-E). The analysis of vaccine efficacy in maternal participants will be based on the Exposed set.

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

# Secondary Efficacy **Statistical Analysis Methods Endpoints** From birth (Visit 1-NB) to 6 months (Visit 4-NB), occurrences of RSV-associated hospitalizations according to the case definitions. From birth (Visit 1-NB) to 6 months (Visit 4-NB), occurrences of all-cause LRTIs From birth (Visit 1-NB) to 6 months (Visit 4-NB), occurrences of all-cause LRTIs with hospitalization From birth (Visit 1-NB) to 12 months, occurrences of severe medically assessed, RSVassociated LRTIs according to the case definitions From birth (Visit 1-NB) to 12 months, occurrences of any medically assessed, RSVassociated LRTIs according to the case definitions. From birth (Visit 1-NB) to 6 months (Visit 4-NB), occurrences of severe medically assessed, RSVassociated LRTIs according to the case definition, for RSV subtype A and RSV subtype B separately. From birth (Visit 1-NB) to 6 months (Visit 4-NB), occurrences of any medically assessed, RSV-associated LRTIs according to the case definition, for RSV subtype A and RSV subtype B separately.

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

| | | Statistical Analysis Plan Amendment 5 |
|---|---|---|
| Secondary Efficacy<br>Endpoints | Statistical Analysis Methods | |
| From birth (Visit 1-NB) to 4 months (Visit 3-NB), occurrences of severe medically assessed, RSV-associated LRTIs according to the case definition. | CCI | |
| From birth (Visit 1-NB) to 4 months (Visit 3-NB), occurrences of any medically assessed, RSV-associated LRTIs according to the case definitions | | |
| From birth (Visit 1-NB) to 6 months (Visit 4-NB), occurrences of all-cause pneumonia | | |
| From study intervention<br>administration (Visit 1) to 6<br>months post-delivery (Contact<br>1), occurrence of RSV-<br>associated medically attended<br>RTIs (RSV-MA-RTIs) | _ | |
| From birth (Visit 1-NB) to 12 months (Visit 5-NB), occurrences of RSV-associated hospitalizations according to the case definitions. | | |

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5



## 5.3. Immunogenicity

## 5.3.1. Analysis of immunogenicity planned in the protocol

All immunogenicity analyses in stage A will be based on the Per Protocol - Immunogenicity set.

Note: In the immunogenicity sub-cohort, only those samples for which a pair (both maternal and respective infant) exist will be analyzed to evaluate secondary immunogenicity objectives and to assess antibody persistence in infants.

When performing experiments to monitor the stability of the RSV NEUT A assay overtime, a QC panel excursion was observed for tests performed after May 2023. Consequently, the testing was temporarily paused and not all samples were tested.

| Secondary Immunogenicity<br>Endpoints – Maternal Participants | Statistical Analysis Methods |
|---|---|
| Neutralizing antibody titers<br>against RSV-A | |
| Measured on blood samples collected at Day 1 before vaccination (Visit 1), at Day 31 (Visit 2), and at delivery (Visit 3). | |
212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

| | Statistical Analysis Flan Amendment 5 |
|---|---|
| Secondary Immunogenicity Endpoints – Cord blood / placental transfer | Statistical Analysis Methods |
| RSVPreF3 IgG-specific antibody concentration measured on blood samples collected at Delivery and cord blood* The ratio between cord blood* and maternal RSVPreF3 IgG- specific antibody concentrations | CCI |
| * or an infant blood sample collected within 72 hours after birth (if no cord blood sample can be obtained). | |
| Secondary Immunogenicity Endpoints – Infant Participants | |
| Neutralizing antibody titers<br>against RSV-A. | |
| Measured on the cord blood sample collected at delivery (or on a blood sample collected from the infant within 72 hours after birth if no cord blood sample can be obtained) and at Day 43 (Visit 2-NB), Day 121 (Visit 3- | |
| NB), or Day 181 (Visit 4-NB) after delivery in 3 sub-cohorts of infants. Infants born to women in the | |
| immunogenicity sub-cohorts will be randomly assigned (1:1:1) to sample collection at 1 of the 3 timepoints noted. | |

## 5.3.2. Additional considerations

## 5.3.2.1. Sensitivity analysis

A sensitivity analysis will be performed based on the Per Protocol-Immunogenicity set excluding participants in Bangladesh.

## 5.3.2.2. Between group analysis





## 5.4. Analysis of safety and reactogenicity

## 5.4.1. Analysis of safety and reactogenicity planned in the protocol

Safety analyses in **maternal participants** will include summaries by study group and age category (18-34, 35-39, ≥40 years of age; overall) of solicited administration site and systemic events (for stage A subjects), unsolicited AEs, MAEs, SAEs, MA-RTIs (RSV-associated MA-RTIs and all-cause MA-RTIs), AEs leading to study withdrawal, pregnancy outcomes and pregnancy related AESIs.

Safety analyses in **infant participants** will include summaries by study group, overall and gestational age at birth (≥ 37 weeks or < 37 weeks) of neonatal AESIs, MAEs, SAEs, AEs leading to study withdrawal, and the occurrence of RSV-associated RTIs, LRTIs, severe LRTIs, RSV-associated hospitalizations, all-cause RTI and all-cause LRTI.

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

Safety analyses for maternal participants and infants may also be reported by economic region (LMIC and HIC).

Analyses of solicited AEs will be performed on the Solicited Safety set (maternal participants only). Analyses of unsolicited AEs will be performed on the ES.

| Primary Safety Endpoints – Infant<br>Participants | Statistical Analysis Methods |
|---|---|
| Occurrence of SAEs, AEs leading to study termination and medically attended AEs from birth up to 6 months after birth | CCI |
| Occurrence of SAEs, AEs leading to study termination and medically attended AEs from birth up to 12 months after birth. | |
| Secondary Safety Endpoints – Maternal Participants | Statistical Analysis Methods |
| Occurrence of solicited injection site and systemic events in Stage A participants during a 7-day follow-up period after vaccination (i.e. the day of vaccination and 6 subsequent days). | CCI |
| Occurrence of unsolicited adverse events (AEs) in all maternal participants during a 30-day follow-up period after vaccination (i.e. the day of vaccination and 29 subsequent days). | |

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

Pregnancy outcomes from Day 1 (Visit 1) up to 6 weeks after delivery (Day 43 post-delivery, Visit 4). These include live birth with no congenital anomalies, live birth with minor congenital anomaly(ies) only; live birth with at least one major congenital anomaly, fetal death/still birth (antepartum or intrapartum) with no congenital anomalies, fetal death/still birth (antepartum or intrapartum) with minor congenital anomalies only, fetal death/still birth (antepartum or intrapartum) with at least 1 major congenital anomaly; elective/therapeutic termination with no congenital anomalies; elective/therapeutic termination with minor congenital anomalies only, and elective/therapeutic termination with at least 1 major congenital anomaly.

Pregnancy-related adverse events (AEs) of special interest from Day 1 (Visit 1) up to 6 weeks after delivery (Day 43 post-delivery, Visit 4). These include maternal death, hypertensive disorders of pregnancy (gestational hypertension, pre-eclampsia, pre-eclampsia with severe features including eclampsia), fetal growth restriction, pathways to preterm birth (premature preterm rupture of membranes, preterm labor, provider-initiated preterm birth), gestational diabetes mellitus, chorioamnionitis.

Occurrence of serious adverse events (SAEs), AEs leading to study termination, and medically attended AEs in all maternal participants from Visit 1 (Day 1) up to 6 months after delivery.

## Secondary Safety Endpoints – Infant Participants

The occurrence of neonatal AEs of special interest (reported up to 6 weeks after birth). These include small for gestational age, low birth weight including very low and extremely low birth weight (<2500 g, <1500g, <1000g), congenital anomalies (major external structural defects, internal structural defects, functional defects), neonatal death (in an extremely preterm birth (22≤GA<28 weeks), in a preterm live birth), preterm birth.

## 5.4.2. Additional considerations

## 5.4.2.1. Analysis of solicited events

The analysis of solicited events will be performed on Solicited Safety Set. The intensity of the following solicited events will be assessed as described:

Table 9 Intensity scales for solicited symptoms in adults

| Adults | | |
|---|---|---|
| Event Intensity grade | | Parameter |
| Pain at administration site | 0 | None |
| | 1 | Mild: Any pain neither interfering with nor preventing normal every day activities. |
| | 2 | Moderate: Painful when limb is moved and interferes with every day activities. |
| | 3 | Severe: Significant pain at rest. Prevents normal every day activities. |
| Redness at administration site | | Record greatest surface diameter in mm |
| Swelling at administration site | | Record greatest surface diameter in mm |
| Temperature* | | Record temperature in °C/°F with 1 decimal Temperature will be analysed in 0.5°C increments from ≥ 38.0°C /100.4°F) Grade 3 fever is defined as > 39.0°C /102.2°F |
| Headache | | |
| Fatigue | 0 | Normal |
| Nausea | 1 | Mild: Easily tolerated |
| Vomiting | 2 | Moderate: Interferes with normal activity |
| Diarrhea | 3 | Severe: Prevents normal activity |
| Abdominal pain | | |

<sup>\*</sup> Preferred location for measurement will be the oral cavity. "Fever" = temperature ≥38.0°C/100.4°F regardless of the location of measurement.

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

The maximum intensity of local injection site (redness and swelling) will be scored at GSK Biologicals as follows:

| 0: | ≤ 20 mm |
|----|--------------------|
| 1: | > 20 mm to ≤50 mm |
| 2: | > 50 mm to ≤100 mm |
| 3: | >100 mm |

Duration in days of solicited administration site and systemic events within 7 days after vaccination will be tabulated by study group and overall, and if needed by age group. The derivation rule of duration in days for solicited events is detailed in section 10.1.2.11.

### 5.4.2.2. Exclusion of implausible solicited Event

Some local and systemic events will be directly measured by the participant and cannot be changed even if they are biologically implausible. Therefore, these implausible measurements will be removed from the analysis but included in listings. Implausible measurements are summarized in the table below:

Table 10 Implausible Solicited Events

| Parameter | Implausible measurements |
|------------------|--------------------------------------|
| Body temperature | ≤ 33°C or ≥ 42°C |
| Erythema | Measurements < 0 mm |
| | For participants ≥ 6 years: ≥ 900 mm |
| Swelling | Measurements < 0 mm |
| | For participants ≥ 6 years: ≥ 500 mm |

## 5.4.2.3. Analysis of Unsolicited Adverse Events

The analysis of unsolicited events will be performed on ES

#### 5.4.2.4. Combined Solicited and Unsolicited Adverse Events

The combined analysis of solicited and unsolicited events will be performed on ES. A summary of participants with all combined solicited and unsolicited adverse events will be provided.

Solicited adverse events will be coded by MedDRA.

For clintrial.gov and EudraCT posting purposes, a summary of combined solicited and unsolicited adverse events will be produced by System Organ Class and preferred terms and according to occurrence of each event.

#### 5.4.2.5. Other analysis

Other safety analysis will be performed on ES.

Concomitant medications will be coded using the GSKDRUG dictionary. The number and percentage of maternal participants taking concomitant medications (any medication, any antipyretic and any antipyretic taken prophylactically, respectively) within 7 days

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

following vaccination, 30 days following vaccination, up to 6 weeks post-delivery and up to 6 months post-delivery will be summarized by group. A listing will also be provided.

The number and percentage of infants taking previous and concomitant medications/vaccinations from birth up to 6 weeks after birth, 6 months after birth and 1 year after birth will be summarized by group. A listing will also be provided.

#### 6. ANALYSIS INTERPRETATION

All comparative analyses will be descriptive with the aim to characterize the difference in immunogenicity between groups. These descriptive analyses should be interpreted with caution considering that there is no adjustment for multiplicity for most of these comparisons.

## 7. CONDUCT OF ANALYSES

## 7.1. Sequence of analyses

An interim analysis of safety endpoints for both maternal and infant participants has been performed, with the focus on demonstrating the safety profile at Day 43 post-delivery. The interim analysis was deemed necessary following the identification of the safety signals documented in protocol amendment 4, which assisted in the better characterization of the safety information including the signals. The interim analysis was performed after all infants completed the 43 days post-delivery timepoint. The safety endpoints are identical to those listed in section 2, and the statistical analysis methods are similar to section 5.4.1. with minor modifications. In addition, summaries of demographics, participant disposition, concomitant medication/vaccinations and medical history was included. This analysis was performed by an external Independent Data Analysis Center (IDAC). In addition, monthly safety analyses are conducted, where most of the analyses have been generated by IDAC and monitored by the SRT on a monthly basis and by an Independent Data Monitoring Committee (IDMC) on a bi-monthly basis. Additional non-standardized ad-hoc analyses (safety signal deep dive) are performed by internal GSK.

6 Month Post-delivery interim analysis occurred as described below:

• When all maternal and infant participants enrolled completed 6 months follow-up post-delivery/birth (to evaluate primary and secondary efficacy endpoints, reactogenicity and safety)

Final analysis will occur as described below:

• When all infant participants have completed Visit 5-NB (month 12, LSLV), a final safety analysis (for all maternal and infant participants in both Stage A and Stage B), a final secondary efficacy analysis up to 12 months follow up post birth, and a final immunogenicity analysis will be performed. Analyses of any evaluated tertiary endpoints may also be performed.

6 Month Post-delivery interim analysis was performed by internal GSK, so will be the final analysis.

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

If the data for tertiary endpoints becomes available at a later stage, (an) additional analysis/analyses will be performed.

| Description | Disclosure Purpose |
|----------------------------------------|---------------------------------|
| Day 43 post-delivery interim analysis | Internal |
| 6 Month post-delivery interim analysis | Public Disclosure. |
| Final Analysis at Month 12 post birth | Public Disclosure, Study Report |

## 7.2. Statistical considerations for interim analyses

Not applicable.

## 8. CHANGES FROM PLANNED ANALYSES

- By-participant listings of SAEs, AEs leading to study withdrawal, MAEs, adverse
  pregnancy outcomes and pregnancy related AESIs will be prepared and released.
  Such listings have already been released in earlier analyses. Due to study
  enrolment/vaccination stop, the study has been unblinded already before the final
  analysis.
- A sensitivity analysis for immunogenicity results excluding participants from Bangladesh, for which HIV testing was not performed before their enrollment into the study, has been added.
- Between group evaluations for immunogenicity analysis was clarified to be performed among RSV MAT and Control instead of vaccination groups, the wording has been corrected.
- In February 2022, enrollment and vaccination were stopped because of an imbalance in preterm births and associated neonatal deaths observed between the RSVPreF3-Mat and placebo groups. Subsequently the study was unblinded, and therefore the presented VE endpoints are descriptive.
- Subgroup analyses by economic region (LMIC and HIC) will be performed for demography, efficacy, and safety evaluations.
- Subgroup analyses by gestational age at birth will be performed for demography and safety evaluations.
- Sensitivity analysis for primary efficacy endpoints by using a negative binominal regression model have been removed.

# 9. NON-STANDARD DATA DERIVATION RULES AND STATISTICAL METHODS

The following sections describe additional derivation rules and statistical methods which are not presented in section 10.1.

## 9.1. Gestational age at vaccination

Gestational age at vaccination in weeks for maternal participants will be entered by the investigator and used for our analyses. It will not be derived from the estimated date of delivery.

## 9.2. Immunogenicity

For a given participant and given immunogenicity measurement, missing or non-evaluable measurements will not be replaced. Therefore, an analysis will exclude participants with missing or non-evaluable measurements.

- For the within-group assessment, the descriptive analysis performed for each assay at each timepoint will exclude participants with a missing or non-evaluable measurement.
- For the between group assessments, statistical model will be fitted based on the participants having a result at both the baseline and the considered timepoint.

The GMT/GMC and its 95% CI will be obtained by exponentiating the mean and its 95% CI of the log-transformed titres/concentrations. All CI computed will be two-sided 95% CI.

Placental transfer is defined as the ratio of RSVPreF3 IgG-specific antibody concentrations between cord blood (or blood sample from infants collected within 3 days after birth if cord blood is not available) and maternal blood sample at delivery (or within 3 days after delivery if blood sample is not collected during delivery).

## 9.2.1. Assay cut-offs

## 9.2.1.1. Assay cut-offs for serology results

A seronegative participant is a participant whose antibody titre is below the cut-off value of the assay. A seropositive participant is a participant whose antibody titre is greater than or equal to the cut-off value of the assay. The cut-off tests for immunogenicity evaluation will be as per following:

| System | Component | Method | Unit | Cut-off<br>(LLOQ) | ULOQ |
|---|---|---|---|---|---|
| Serum | RSV-A Neutralising Antibody | CCI | | | |
| Serum | RSVPreF3 IgG antibody concentrations | | | | |
| Serum | RSV-B Neutralising Antibody* | | | | |

Note: the assay cut-off (LLOQ), ULOQ and units may be further adjusted at time of analysis.

## 9.2.1.1.1. Assay cut-offs for central nasal swabs

| System | Component | Method | Unit | Cut-off |
|------------|----------------|--------|------|---------|
| Nasal Swab | RSV-A positive | CCI | | |
| Nasal Swab | RSV-B positive | | | |

<sup>\*:</sup> RSV-B neutralizing antibody titers will no longer be assessed as part of the secondary immunogenicity endpoints.

### 9.2.2. RTI and LRTI

Cases will be classified (during data analyses) according to the definitions that follow.

Table 11 MA-RTI case definitions for data analysis in maternal participants

| RSV-MA-RTI | Medically attended visit for RTI symptoms AND Confirmed RSV infection <sup>1, 2</sup> |
|---|---|
| RSV hospitalization | Confirmed RSV infection AND |
| | Hospitalized for acute medical condition <sup>3</sup> |
| All-cause MA- RTI | Medically attended visit for RTI symptoms |

<sup>&</sup>lt;sup>1</sup> Confirmed RSV infection defined in Section 4.2.6.3 of the Protocol

MA-RTI = Maternal, medically attended respiratory tract illness

Table 12 RTI/LRTI case definitions for data analysis in infants

| RSV-RTI | Runny nose, <b>OR</b> Blocked nose, <b>OR</b> Cough |
|---|---|
| | AND |
| | Confirmed RSV infection 4,5 |
| RSV-LRTI | History of cough <b>OR</b> difficulty in breathing <sup>1</sup> |
| | AND |
| | SpO <sub>2</sub> < 95% <sup>2</sup> , <b>OR</b> RR increase <sup>3</sup> |
| | AND |
| | Confirmed RSV infection 4,5 |
| RSV-severe LRTI | Meeting the case definition of RSV-LRTI |
| | AND |
| | SpO <sub>2</sub> < 93% <sup>2</sup> , OR lower chest wall in-drawing <b>OR</b> inability to feed <b>OR</b> failure to |
| | respond/unconscious |
| RSV hospitalization | Confirmed RSV infection 4,5 |
| | AND |
| | Hospitalized for acute medical condition <sup>6</sup> |
| All-cause RTI | Runny nose, OR Blocked nose, OR Cough |
| All-cause LRTI | History of cough <b>OR</b> difficulty in breathing <sup>1</sup> |
| | AND |
| | SpO2 < 95% <sup>2</sup> , <b>OR</b> RR increase <sup>3</sup> |
| All-cause LRTI hospitalization | Hospitalized due to all cause LRTI as defined above |

Definitions based on [Modjarrad, 2016]; except that definitions for severe and very severe RSV LRTI have been merged. **RTI** = respiratory tract illness; **LRTI** = lower respiratory tract illness; **RR** = respiratory rate; **SpO**<sub>2</sub> = blood oxygen saturation by pulse oximetry.

- > 60/minute (< 2 months of age)
- > 50/minute (2 to < 12 months of age)
- > 40/minute (12 to 24 months of age)
- <sup>4</sup> Confirmed RSV infection
- <sup>5</sup> RSV (nasal swab) sampling and testing

<sup>&</sup>lt;sup>2</sup> RSV (nasal swab) sampling and testing as specified in Table 14 of the Protocol.

<sup>&</sup>lt;sup>3</sup> Hospitalization is defined as admission for observation or treatment based on the judgement of a health care provider.

<sup>&</sup>lt;sup>1</sup> Based on history reported by parents/LARs and includes difficulty in breathing (e.g. showing signs of wheezing or stridor, tachypnoea, flaring [of nostrils], chest in-drawing, apnea).

<sup>&</sup>lt;sup>2</sup> For blood oxygen saturation (SpO<sub>2</sub>), the lowest value monitored will be used. In high altitudes (>2500m), SpO<sub>2</sub> <92% for LRTI, <90% for severe LRTI.

<sup>&</sup>lt;sup>3</sup> RR increase defined as:

<sup>&</sup>lt;sup>6</sup> Hospitalization is defined as admission for observation or treatment based on the judgement of a health care provider.

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

For RSV infection the sponsor will analyse nasal swabs by quantitative reverse transcription polymerase chain reaction (qRT-PCR) for the presence of RSV A/B. A positive (RSV A or B) test result constitutes a case of RSV infection.

In the event the collection of a nasal swab for testing by the sponsor is impossible, results from locally collected samples, tested with locally approved tests, may also be considered for the determination of a case of RSV infection.

For the analysis of RTI episode, a new RTI episode will be defined as any occurrence of cough and/or difficulty in breathing with an interval of at least 7 consecutive days without cough and/or difficulty in breathing since the last/previous episode of RTI.

## 9.2.2.1. Alternative LRTI / Severe LRTI case definitions for data analysis in infants

To meet an alternative case definition, a participant must have at least one item from each column.

Note: As per protocol amendment 5, the alternative case definitions will no longer be considered for data analysis in infants.

Table 13 Alternative LRTI / Severe LRTI case definitions in infants

| | RSV confirmed | Documented PE findings indicating lower respiratory tract involvement | Objective measures of clinical severity |
|---|---|---|---|
| LRTI | Confirmed RSV infection | Rhonchi<br>Crackles (Rales)<br>Wheeze | Increased respiratory rate (bpm) ■ ≥ 60 for < 2 mo ■ ≥ 50 for 2-6 mo Hypoxemia ■ SpO2 <95% at ≤1800 meters ■ SpO2 <92% at > 1800 meters New onset apnea Nasal flaring Retractions Grunting |
| Severe LRTI | Confirmed RSV infection | Rhonchi<br>Crackles (Rales)<br>Wheeze | Hypoxemia ■ Sp02 <93% at ≤1800 meters ■ Sp02 <90% at > 1800 meters Acute hypoxic or ventilatory failure Dehydration due to respiratory distress requiring IV hydration Failure to respond or unconscious |

## 9.2.3. Hematology and Biochemistry parameters

In order to assess the impact of fluid shifts on the antibody concentration/titer, hematocrit will be evaluated at all three blood sampling timepoints (Day 1, Day 31, and delivery) for a subset of maternal (Stage A) participants in the immunogenicity sub-cohort, if deemed necessary.

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

Note that hematocrit sample collection will end once Protocol Amendment 2 becomes effective in the different countries/sites.

## 9.3. Statistical Method

Study Specific statistical methods for immunogenicity analysis are described in section 5.3.

## 10. ANNEXES

# 10.1. Business rules for standard data derivations and statistical methods

This section contains GSK Vaccines' standard rules for data display and derivation for clinical and epidemiological studies. These rules will be applied along with those detailed in section 9 (additional study-specific rules).

## 10.1.1. Handling of missing data





#### 10.1.2. Data derivation

## 10.1.2.1. Age at vaccination in days

When age at vaccination is to be displayed in days, it will be calculated as:

Age = date of vaccination minus date of birth

#### 10.1.2.2. Age at vaccination in months

When age at vaccination is to be displayed in months, it will be calculated as the number of complete calendar months between the date of birth (DOB) and the date of vaccination. For example:

DOB = 10JUN2017, Date of vaccination = 09JUL2018 -> Age = 12 months DOB = 10JUN2017, Date of vaccination = 10JUL2018 -> Age = 13 months

## 10.1.2.3. Age at vaccination in years

When age at vaccination is to be displayed in years, it will be calculated as the number of complete calendar years between the date of birth and the date of vaccination. For example:

DOB = 10SEP1983, Date of vaccination = 09SEP2018 -> Age = 34 years

DOB = 10SEP1983, Date of vaccination = 10SEP2018 -> Age = 35 years

## 10.1.2.4. Weight

Weight will be presented in kilograms or grams. Weights reported in pounds will be converted as follows:

Weight in kilograms = Weight in pounds / 2.2

Weight in grams = (Weight in pound / 2.2)  $\cdot 1000$ 

### 10.1.2.5. Height/Length

Height/Length will be presented in centimeters. Heights/Lengths reported in feet and inches will be converted as follows:

Height/Length in centimeters = Height/Length in inches  $\times 2.54$ 

## 10.1.2.6. Body mass index (BMI)

BMI will be calculated as follows:

BMI = (Weight in kilograms) / (Height in meters)2

## 10.1.2.7. Temperature

Temperatures will be presented in degrees Celsius (°C). Temperatures reported in degrees Fahrenheit (°F) will be converted as follows:

Temperature (Celsius) =  $((Temperature (Fahrenheit) - 32) \times 5)/9$ 

#### 10.1.2.8. Numerical serology results

Numerical serology results will be derived from the content of IS.ISORRES in the SDTM dataset. For assays with a specific cut-off, the following derivation rules apply:

| IS.ISORRES | Derived value |
|-----------------------------------------|---------------|
| "NEG", "-", or "(-)" | cut-off/2 |
| "POS", "+", or "(+)" | cut-off |
| "< value" and value is <= assay cut-off | cut-off/2 |
| "< value" and value is > assay cut-off | Value |
| "> value" and value is < assay cut-off | cut-off/2 |
| "> value" and value is >= assay cut-off | Value |
| "value" and value is < cut-off | cut-off/2 |
| "value" and value is >= cut-off | Value |
| All other cases | Missing |

## 10.1.2.9. Geometric mean titres (GMTs) and concentrations (GMCs)

Geometric Mean Titre (GMT) or Concentration (GMC) calculations are performed by taking the inverse logarithm of the mean of the log titre or concentration transformations. Non quantifiable antibody titres or concentrations will be converted as described in

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

section 10.1.2.8 for the purpose of GMT/GMC calculation. Cut-off values are defined by the laboratory before the analysis.

## 10.1.2.10. Onset day

The onset day for an event (e.g. AE, medication, vaccination) is the number of days between study vaccination and the start date of the event. This is 1 for an event occurring on the same day as vaccination (and reported as starting after vaccination).

The onset day for an event (e.g. neonatal AEs, SAEs, AEs of special interest) for infants is the number of days between birth and the start date of the event (or date of diagnosis). This is 1 for an event occurring on the same day as birth.

#### 10.1.2.11. Duration of events

The duration of an event with a start and end date will be the number of days between the start and end dates plus one day, i.e. an event that starts on 03MAR2018 and ends on 12MAR2018 has a duration of 10 days.

The duration of solicited events will be calculated as the sum of the individual days with the adverse event reported at grade 1 or higher during the solicited adverse event period.

## 10.1.2.12. Counting rules for combining solicited and unsolicited adverse events

For output combining solicited and unsolicited adverse events, all serious adverse events will be considered systemic events since the administration site flag is not included in the expedited adverse event CRF pages. Unsolicited adverse events with missing administration site flag will also be considered systemic.

Multiple events with the same preferred term which start on the same day are counted as only one occurrence.

#### 10.1.2.13. Counting rules for occurrences of solicited adverse events

When the occurrences of solicited adverse events are summarized, each event recorded as having occurred during a specific period will be counted as only one occurrence regardless of the number of days on which it occurs. Also, in the case of co-administered study vaccines, an injection site reaction recorded for a participant following multiple vaccines will be counted as only one occurrence.

## 10.1.3. Display of decimals

### 10.1.3.1. Percentages

Percentages and their corresponding confidence limits will be displayed with one decimal except for 100% in which case no decimal will be displayed.

### 10.1.3.2. Differences in percentages

Differences in percentages and their corresponding confidence limits will be displayed with two decimals.

### 10.1.3.3. Demographic/baseline characteristics statistics

The mean, median, and standard deviation for continuous baseline characteristics (height, weight, body mass index (BMI), pre-vaccination body temperature) will be presented with one decimal.

The minimum and maximum values and quartile values (if required) will be presented with the same number of decimals as the observed values.

The maxima and minima of transformed height/<u>length/weight</u> variables will be displayed without decimals, with the exception of infant studies where three decimals will be displayed for transformed birth weight.

The maximum and minimum of transformed body temperatures will be displayed with one decimal.

## 10.1.3.4. Serological summary statistics

The number of decimals used when displaying geometric mean titers (GMT) or concentrations (GMC) and their confidence limits is assay specific based on the magnitude of the assay result post-dose and the clinically relevant assay threshold. The same number of decimals will be used for a given assay regardless of the timepoint presented.

| Lowest clinically relevant threshold | Example | Number of decimals to display |
|---|---|---|
| < 0.3 | Diphtheria, tetanus, anti-PRP | 3 |
| >=0.3 and <4 | Streptococcus pneumoniae, Meningococal bactericide | 2 |
| >=4 and <1000 | Measles, rubella, varicella, | 1 |
| >=1000 | CMI | 0 |

GMT/GMC fold increase from pre-dose follows the same principle. Namely when the lowest clinically relevant threshold is 2 fold, 2 decimals are displayed while when the lowest clinically relevant threshold is 4 fold, 1 decimal is displayed.

GMT or GMC group ratios and their confidence limits will be displayed with 2 decimals regardless of the actual values.

## 10.1.4. Statistical methodology

### 10.1.4.1. Exact confidence intervals around proportions

The exact confidence intervals around within-group proportions are derived using the method of Clopper and Pearson [Clopper, 1934].

## 10.1.4.2. Standardized asymptotic confidence intervals around differences in proportions

The standardized asymptotic confidence intervals around differences in proportions are derived using the method of Miettinen and Nurminen [Miettinen, 1985]

## 10.1.4.3. Adjusted GMT or GMC ratios

The CI for GMC ratio and adjusted CMT will be obtained using an ANOVA model on the logarithm transformed titers. The ANOVA model will include the vaccine group as the fixed effect (3 groups) and the country effect. The GMC ratio and their 95% CI will be derived by exponential transformation of the corresponding group contrast in the model.

When between-group GMT or GMC ratios are computed and adjusted for two-level categorical co-variables, these co-variables should be included as dummy continuous variables in the SAS procedure. It should also be clear whether the model is limited to the data from some groups.

## 10.2. TFL TOC

The Table Figure Listing (TFL) TOC which itemizes the planned list of TFL and their associated lay-out is developed as a separate document. There will be one TOC document for the interim analysis of Day43PD and another for the 6-month PD interim analysis and the final analysis.

212171 (RSV MAT-009) Statistical Analysis Plan Amendment 5

## 11. REFERENCES

Clopper CJ, Pearson E. The Use of Confidence or Fiducial Limits Illustrated in the case of the Binomial. *Biometrika*. 1934; 26:404-13.

Miettinen, O.S. and Nurminen, M. Comparative analysis of two rates. *Statistics in Medicine*, 1985; 4: 213-226.

Modjarrad K, Giersing B, Kaslow DC, Smith PG, Moorthy VS; WHO RSV Vaccine Consultation Expert Group. WHO consultation on Respiratory Syncytial Virus Vaccine Development Report from a World Health Organization Meeting held on 23-24 March 2015. Vaccine. 2016; 34(2):190-7.